CLINICAL TRIAL: NCT03310034
Title: The Effects of NAD+-Precursor Supplementation on Energy Metabolism in Physically Compromised Elderly
Brief Title: NAD Supplementation Study
Acronym: NADS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Concluded study following COVID19 outbreak and inability to complete study as designed.
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, Patrick Schrauwen, Prof. Dr. P. Schrauwen, Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL61204.068.17
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-03

CONDITIONS: Aging; Mitochondrial Function

STUDY DESIGN:
Intervention Model Description: Randomized, dubbel-blind, cross-over trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Dietary Supplement: NAD-precursors
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: NAD-precursors — Intervention product containing the NAD+-precursors nicotinic acid, nicotinamide, and tryptophan (total of 204 NE per serving) in a whey protein source for 31 days.
  Arms: Intervention
Dietary Supplement: Control — Control product containing amino-acid mixture resembling whey-protein not containing the NAD+-precursors nicotinic acid, nicotinamide, and tryptophan. To be taken for 31 days.
  Arms: Control

SUMMARY:
This research project aims to determine whether supplementing with a mixture of the NAD+-precursors NA, NAM, and tryptophan can stimulate skeletal muscle mitochondrial function in physically compromised, elderly humans. Outcomes are related to mitochondrial function, energy metabolism, and physical function will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age ≥ 65 ≤ 75 years;
* BMI ≥ 20 kg/m2 ≤ 30 kg/m2;
* Normal physical activity levels: maximum of 1 hour per week engagement in a structured exercise session;
* SPPB score 4-9 and (pre-)frail;
* Subject should be in sufficient health to participate in the experiments, to be judged by the responsible physician based on the subject's medical history.

Exclusion Criteria:

* Not meeting all inclusion criteria;
* Smoking;
* Excessive alcohol use and/or drug abuse;
* Subjects with diabetes mellitus type 2;
* Significant food allergies or intolerances concerning the study products;
* Participation in another biomedical study within 1 month before the first study visit, possibly interfering with the study results;
* Medication use known to hamper subject's safety during the study procedures;
* Subjects who use selective serotonin re-uptake inhibitors (SSRI), or selective norepinephrin re-uptake inhibitors (SNRI), or monoamino oxidase inhibitors (MAO-inhibitors), or clomipramine, or St. John's wort (Hypericum perforatum);
* Subjects with contra-indications for MRI;
* Subjects who do not want to be informed about unexpected medical findings;
* Subjects who do not want that their treating physician to be informed;
* Co-morbidities to which the intervention or program the may pose as a complicating factor;
* Inability to participate and/or complete the required measurements.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Ex vivo mitochondrial respiration | After 4 weeks of supplementation.
  Ex vivo mitochondrial function in skeletal muscle measured by oxygen consumption in muscle fibres (muscle biopsy vastus lateralis) on lipid-derived and carbohydrate-derived substrates.
Basal metabolic rate | After 4 weeks of supplementation.
  Basal metabolic rate expressed as kcal/kg/min
In vivo mitochondrial capacity | After 4 weeks of supplementation.
  In vivo mitochondrial capacity measured with 31P-MRS.
Submaximal exercise energy expenditure | After 4 weeks of supplementation.
  Submaximal exercise energy expenditure expressed as kcal/kg/min

SECONDARY OUTCOMES:
Glucose tolerance | After 4 weeks of supplementation.
  Glucose tolerance measured by oral glucose tolerance test.
Ectopic lipid accumulation | After 4 weeks of supplementation.
  Liver and skeletal muscle lipid accumulation measured with H-MRS in vivo.
Acetylcarnitine levels | After 4 weeks of supplementation.
  Skeletal muscle acetylcarnitine levels measured with H-MRS in vivo, before and after exercise stimulation (cycling).
Physical function | After 4 weeks of supplementation.
  Measured by Short Physical Performance Battery and Frailty criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Connell NJ, Grevendonk L, Fealy CE, Moonen-Kornips E, Bruls YMH, Schrauwen-Hinderling VB, de Vogel J, Hageman R, Geurts J, Zapata-Perez R, Houtkooper RH, Havekes B, Hoeks J, Schrauwen P. NAD+-Precursor Supplementation With L-Tryptophan, Nicotinic Acid, and Nicotinamide Does Not Affect Mitochondrial Function or Skeletal Muscle Function in Physically Compromised Older Adults. J Nutr. 2021 Oct 1;151(10):2917-2931. doi: 10.1093/jn/nxab193. PMID 34191033